CLINICAL TRIAL: NCT03528265
Title: Adapting a Rapid Lateral Flow Burkholderia Pseudomallei Immunoassay in Sarawak, Malaysia
Brief Title: Adapting LFI for Melioidosis
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00091842
Record Dates: First submitted 2018-05-07; First posted 2018-05-17 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2018-07

CONDITIONS: Melioidosis
Keywords: lateral flow immunoassay; validation
MeSH Terms: conditions — Melioidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA from blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients with melioidosis-like symptoms admitted to Kapit Hosp
  Interventions: Device: Lateral flow immunoassay

INTERVENTIONS:
Device: Lateral flow immunoassay — Biospecimens of patients with melioidosis-like symptoms will be tested with lateral flow immunoassay to detect Burkholderia pseudomallei, bacterium causing melioidosis

SUMMARY:
Towards the goal of reducing melioidosis, this study will help clinicians in Sarawak to diagnose and understand the causes and risk factors for melioidosis. The data will help the clinicians to provide faster test results and better clinical care. The investigator's laboratory efforts will supplement available diagnostics by adding a new, easier-to-use test involving lateral flow immunoassay to rapidly detect Burkholderia pseudomallei, a bacterium causing melioidosis. The study aims to study up to 400 patients with melioidosis-like symptoms who are admitted to Kapit Hospital, Sarawak, Malaysia. No participants will be enrolled from other sites. The study will also examine the demographic, behavioral and occupational risk factors associated with hospital admissions to understand any existing associations between these variables and melioidosis prevalence.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Kapit Hospital
* Fever more than 3 days and one or more of the following:

  * Enlarged cervical, inguinal or axillary lymph nodes (greater than 3 cm in diameter), painless adenopathy or lymphadenitis or lymph node abscesses
  * One or both sides glands involvement such as tender swelling over medial aspect of the lower eyelid of the lacrimal glands; submandibular glands, parotic glands
  * Bedside scan with splenic or liver hypoechoic lesion (less than 2cm in diameter)
  * Pneumonia not responding to 48 hours of first line antibiotics
  * One or more joint pain with swelling
  * Purplish vesicle or bullae mainly over the lower limbs, may resulting in ulcer after rupture
  * Deep seated abscess or brain abscess or genitourinary abscess or osteomyelitis
  * Severe sepsis patient with or without shock and/or with multiorgan involvement

Exclusion Criteria:

* Have a clear alternative diagnosis other than melioidosis by a trained health care professional at the Kapit Hospital
* Have already been treated for melioidosis (e.g. received antibiotics before the start of the study)
* Are younger than 6 months of age

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients evaluated at Kapit Hospital experiencing melioidosis-like symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Proportion of true positive | up to 5 weeks
  Proportion of true positive of Bukholderia pseudomallei using rapid diagnostic tests compared to the results of qPCR, bacterial culture and Gram stain
Proportion of true negative | up to 5 weeks
  Proportion of true negative of Bukholderia pseudomallei using rapid diagnostic tests compared to the results of qPCR, bacterial culture and Gram stain

SECONDARY OUTCOMES:
Statistical association between risk factors and test results | up to 3 months
  conduct a survey to determine a statistical association between clinical risk factors and the test results combined

CONTACTS AND LOCATIONS:
Overall Officials: Gregory C Gray, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Kapit Hospital, Kapit, Sarawak, Malaysia

IPD SHARING:
Plan to Share IPD: No